CLINICAL TRIAL: NCT06905925
Title: The Effect of the Training Program Given to Permanent Colostomy Patients on Self-efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cansel Bozer, lecturer, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-03
Record Dates: First submitted 2024-12-08; First posted 2025-04-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stoma Colostomy; Colo-rectal Cancer
Keywords: stoma; Colo-rectal cancer; consulting; self-efficacy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: To eliminate selection bias and ensure balance in the number of patients between groups, randomization will be performed in the study. Randomization will be generated by an independent researcher not involved in the study using a computer tool (https://www.randomizer.org/), and X envelopes will be numbered from 1 to X. Inside the envelopes, cards will indicate whether the participant belongs to the intervention or control group based on the randomization table. Participants who are admitted to the clinic and consent to participate in the study by signing the consent form will be assigned to the intervention or control group based on the envelope number corresponding to their admission order. Once the researcher obtains written consent from the participants, they will open the envelope to determine which group the participant belongs to. This process ensures that randomization and group assignment are concealed, thus controlling for selection bias in the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Written consent will be obtained from the patients in both the intervention and control groups one day before or on the day of surgery. A "Personal Information Form" will be completed through face-to-face interviews with patients who agree to participate in the study. This process is expected to take approximately 5 minutes.
  Patients in the experimental group will receive pre-operative stoma care education from the researcher. This training is expected to last about 15 minutes. After the training, a brochure will be provided to the patients that they can use if they need further information. During the training process, patients will be informed that the researcher will contact them by phone after discharge during the 1st, 2nd, 3rd, and 4th weeks. During these calls, patients will be asked weekly (during weeks 1, 2, 3, and 4) about the color, odor, texture of the wound area, the function of the colostomy, and any complications. In addition, at the end of the 2nd week, if there are no
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no intervention group (No Intervention): No intervention will be performed by the researcher for the patients in the control group. During this process, standard care education will be provided by clinical nurses, and phone follow-up and counseling protocols will not be applied. Patients in the control group will also be contacted by phone by the researcher during the 2nd and 4th weeks after discharge to complete the "Stoma Self-Efficacy Scale (S-SES)."
- intervention group (Experimental): Here is the English translation of the provided text:
  Patients in the experimental group will receive pre-operative stoma care education from the researcher. This training is expected to last approximately 15 minutes. After the training, a brochure will be provided to the patients, which they can use if they need additional information. During the training process, patients will be informed that the researcher will contact them by phone during the 1st, 2nd, 3rd, and 4th weeks after discharge. During these calls, patients will be asked weekly (during weeks 1, 2, 3, and 4) about the color, odor, texture of the wound area, the function of the colostomy, and any complications. Additionally, at the end of the 2nd week, if there are no issues around the wound or sutures, patients will be called to the hospital for suture removal and dressing changes. In other weeks, dietary habits and the condition of the wound will also be inquired. During this four-week period, patients or their relativ
  Interventions: Other: The group receiving counseling

INTERVENTIONS:
Other: The group receiving counseling — Patients in the experimental group will receive pre-operative stoma care education from the researcher. This training is expected to last approximately 15 minutes. After the training, a brochure will be provided to the patients, which they can use if they need additional information. During the training process, patients will be informed that the researcher will contact them by phone during the 1st, 2nd, 3rd, and 4th weeks after discharge. During these calls, patients will be asked weekly (during weeks 1, 2, 3, and 4) about the color, odor, texture of the wound area, the function of the colostomy, and any complications. Additionally, at the end of the 2nd week, if there are no issues around the wound or sutures, patients will be called to the hospital for suture removal and dressing changes. In other weeks, dietary habits and the condition of the wound will also be inquired. During this four-week period, patients or their relatives will be informed that they can contact the researcher
  Arms: intervention group

SUMMARY:
The planned research aims to evaluate the impact of a training program on self-efficacy in patients with permanent colostomies. It highlights the importance of holistic patient education in preventing complications and improving adaptation to stomas, which can positively affect patients' quality of life and self-efficacy.

DETAILED DESCRIPTION:
Stomas can be either temporary or permanent. Stomas can cause physical issues such as uncontrolled gas output, bad odor, leakage, and local skin irritation, as well as psychological and social problems such as sexual dysfunction, changes in body image, decreased self-esteem, interpersonal relationship issues, depression, anxiety, loneliness, fear, and shame. These problems can reduce individuals' self-care abilities, negatively affect daily living activities, increase their vulnerability to stoma/peristomal complications, and further delay the closure of temporary stomas. Regardless of the type of stoma, all of these issues negatively impact patients' self-efficacy.

Many of these problems and potential complications after stoma formation are preventable. Patient education provided through a holistic approach covering pre-operative, post-operative, and home care and follow-up is of great importance in preventing complications and improving patients' adaptation to the stoma. However, a review of the literature reveals that stoma-related education programs typically focus on assessing quality of life and similar factors. Some of the studies reviewed include educational content on pre-operative patient preparation and post-operative care, while others focus only on post-operative complication management. However, high-evidence guidelines, such as Enhanced Recovery After Surgery (ERAS) protocols, emphasize that the first step toward a successful surgical process should be patient education delivered through a holistic approach covering the entire surgical process.

Therefore, the planned research will be conducted to evaluate the effect of a training program provided to patients with permanent colostomies on self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* • Patients scheduled for permanent colostomy following colorectal surgery,

  * Aged 18 years and older,
  * Conscious, with orientation to person, time, and place,
  * Able to speak Turkish,
  * Without auditory or visual impairments,
  * Using a phone, were included in the study. Exclusion Criteria:• Patients who could not be contacted during the study period, or those who developed post-operative complications (such as stenosis, necrosis, ileus, dermatitis, parastomal herniation, etc.) were excluded from the sample.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Stoma Self-Efficacy Scale (S-SES) | 1 years
  The scale was developed to examine the self-efficacy status of patients with stoma. Its validity and reliability in Turkish were conducted by Karaçay et al. The scale consists of 22 items and two subscales. The scale is a 5-point Kickert type, rated from 1 to 5, where 1: definitely do not trust and 5: definitely trust. Items 1-13 of the scale examine Stoma Care Self-Efficacy (S-SES Care), and items 14-22 examine Social Life Self-Efficacy (S-SES Social). The lowest score that can be obtained from the scale is 22, while the highest score is 110. A higher score indicates higher self-efficacy. In the Turkish validity-reliability study of the scale, the Croncbach alpha coefficient was found to be 0.95

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to for personal reasons.